CLINICAL TRIAL: NCT06508372
Title: Efficacy and Safety of Thymoquinone Ointment as a Potential New Therapeutic Modality of Psoriasis Vulgaris.
Brief Title: Topical Thymoquinone in Psoriasis Vulgaris
Status: Not yet recruiting | Phase: Not Applicable | Type: Interventional
Sponsor: Assiut University (Other)
Responsible Party: Principal Investigator, Heba Hasan Sayed, Doctor, Assiut University
Allocation: Randomized | Model: Single Group | Masking: Triple | Purpose: Treatment
Other Study IDs: Topical thymoquinone
Record Dates: First submitted 2024-07-08; First posted 2024-07-18 (Actual); Last update posted 2024-07-19 (Actual); Status verified 2024-07

CONDITIONS: Psoriasis Vulgaris
Keywords: topical thymoquinone

STUDY DESIGN:
Intervention Model Description: Intrapatient randomized controlled study: Topical Thymoquinone ointment will be applied to one psoriatic plaque on one side of the body, while the placebo ointment will be applied to a similar psoriatic plaque on the other side of the body twice daily for 3 months. each patient is randomizied to receive topical thymoquinone ointment on either the left or the right side.
Who Masked: Participant, Care Provider, Investigator
Oversight: FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (2):
- topical thymoquinone ointment (Experimental): One plaque on one side of the body per every patient will be selected, whose diameter would not exceed 5-10 cm2 to apply Thymoquinone ointment as a monotherapeutic ttt twice daily for 3 months.
  Interventions: Drug: Topical thymoquinone Ointment
- topical placebo ointment (Placebo Comparator): In each patient a single similar psoriatic plaque on the other side of the body [as regard anatomical site, size and TES (thickness, erythema, scales) score] will be treated with placebo ointment twice daily for 3 months as a control.
  Interventions: Drug: topical placebo ointment

INTERVENTIONS:
Drug: Topical thymoquinone Ointment — One plaque per patient on one side of the body will be selected, whose diameter would not exceed 5-10 cm2 to apply Thymoquinone ointment as a monotherapeutic ttt twice daily for 3 months.
  Arms: topical thymoquinone ointment
Drug: topical placebo ointment — In each patient a single similar psoriatic plaque on the other side of the body [as regard anatomical site, size and TES (thickness, erythema, scales) score] will be treated with placebo ointment twice daily for 3 months as a control.
  Arms: topical placebo ointment

SUMMARY:
A previous trial found that N. sativa oil was more effective as an antipsoriatic agent, particularly when taken as both a cream and a pill. This confirmed that N. sativa possesses antipsoriatic properties and can alleviate psoriasis symptoms

DETAILED DESCRIPTION:
Psoriasis is a systemic chronic relapsing immune-mediated disease which often requires a long-term therapy. Psoriasis occurs in around 2-3% of the total global population. In Egypt, the prevalence of psoriasis ranges between 0.19% and 3%.

Besides, it could have profound implications on the patients' psychological state and quality of life.

It is presented by erythematous, scaly plaques over the preferred sites. The pathogenesis of this highly complex disease is still far from being fully understood. Keratinocytes' hyperproliferation and immune system dysfunctions are well recognized contributors, with numerous treatments targeting these unique immunologic dysfunctions.

Topical therapy for psoriasis is a current trending subject as it implies good compliance for the patient, few adverse systemic reactions and a targeted effect. Numerous substances are now being tested, from natural to synthetic compounds and already known substances in improved formulas such as vesicular systems.

Nigella sativa belongs to the Ranunculaceae family is an annual plant which distributed in southern Europe and some parts of Asia, including Syria, Turkey, Saudi Arabia, Pakistan, and India. Different active pharmaceutical ingredients have been identified in the N. sativa seeds, including saponins, flavonoids, cardiac glycosides, thymoquinone, thymol, limonene, carvacrol, p-cymene, alpha-pinene, 4-terpineol, longifolene, t-anethole benzene, isoquinoline, and pyrazole alkaloids, as well as unsaturated fatty acid such as linoleic acid, oleic acid, and palmitic acid.

Thymoquinone is the major bioactive ingredient, accounting for 30-48% of the essential oil, has high antioxidant and anti-inflammatory, immune-boosting, cell survival-improving, and energy metabolism-promoting properties, which may explain why they are so beneficial to our health. The anti-inflammatory properties of black seeds and thymoquinone are primarily mediated by COX-2 and PGD2 inhibition.

Clinical trials on skin disorders have shown that N. sativa essential oil and crude extract are effective. (Atopic dermatitis, Atopic eczema,Wart, Eczema, Acne vulgaris, Acute cutaneous leshmaniasis, Arsenical keratosis, Psoriasis, Vitiligo, Infant skin infections, Acute radiation dermatitis) It can be applied as an alternative treatment that helps patients with skin-related problems

ELIGIBILITY:
Inclusion Criteria:

* Patients with clinical diagnosis of mild psoriasis vulgaris
* Age: between 18 and 60 years' old
* Patients who stopped any systemic therapy or phototherapy for at least 3 months and topical therapy for at least 4 weeks prior to enrollment

Exclusion Criteria:

* Psoriasis vulgaris involving > 10% of the body surface area, pustular or erythrodermic psoriasis.
* Pregnant or lactating females.
* Patients with any current dermatological disease.
* Patients with any current systemic disease.

Ages: 18 Years to 60 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult
Enrollment: 30 (Estimated)
Dates: Start 2024-08-01 (Estimated); Primary Completion 2024-12 (Estimated); Study Completion 2025-01 (Estimated)

PRIMARY OUTCOMES:
Psoriasis severity score (TES) assessment | 3 months
  Psoriasis severity score (TES): It is a physician-based, four-point scoring system in which the thickness, erythema, and scales within each plaque will be rated from 0 (none) to 3 (severe)at baseline and to evaluate the therapeutic outcome of topical thymoquinone ointment in each follow up visit.

SECONDARY OUTCOMES:
Evaluation of treatment adverse effects | 3 months
  Any local or systemic side effects will be reported to evaluate the safety of Thymoquinone ointment for treatment of localized plaque psoriasis

IPD SHARING:
Plan to Share IPD: No

REFERENCES:
- [Background] Omar SS, Helaly HA. Prevalence of ocular findings in a sample of Egyptian patients with psoriasis. Indian J Dermatol Venereol Leprol. 2018 Jan-Feb;84(1):34-38. doi: 10.4103/ijdvl.IJDVL_1239_15. PMID 29067934